CLINICAL TRIAL: NCT00485446
Title: Thrombophilia and Thyroid Autoimmunity in Implantation Failure and Recurrent Miscarriage
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Other Study IDs: VLC-JB-0304-307-10
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Thrombophilia, Thyroid Autoimmunity
MeSH Terms: conditions — Thrombophilia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: blood analysis

SUMMARY:
This study was designed to evaluate the incidence of both, inherited and adquired thrombophilia, and thyroid autoinmunity in unknown infertility (UI), implantation failure (IF) and recurrent miscarriage (RM). To focus on these particular disorders and to rule out another potential confounding variables, 4 particular groups of women were created. Only young women (< 38 years old), patients whose previous preimplantation genetic screening (PGS) cycles displayed an acceptable rate of aneploidies, and women without organic uterine abnormality, autoimmune disease or endocrine disorder were included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. The control group included 32 oocyte donors, 18-35 years old, white caucasian, with normal karyotype, no miscarriages, and previous healthy live born infants without pregnancy complications.
2. The UI group consisted of 31 couples with > 1 year infertility , < 38 years of age, normal ovarian function, normal hysterosalpingography and transvaginal ultrasound scan of the uterus and ovaries, normal karyotype in both parents, and normozoospermia.
3. The IF group included 26 couples with 3.9±1.1 IVF failures with embryo transfer of at least 2 good quality embryos. They were < 38 years old, white caucasian, and had normal uterus by vaginal ultrasound and/or hysterosalpingography/ hysteroscopy. Moreover, endocrine disorders or autoimmune diseases were ruled out, a normal karyotype was found in both parents. The male had a sperm concentration > 5 mill/ml.They also had a PGS cycle with ≥ 60% of normal embryos.
4. The group of women with RM (n = 30) had 3.2±1.3 (range: 2-9) previous miscarriages. They were < 38 years old, white caucasian, with normal uterus by vaginal ultrasound and/or hysterosalpingography/ hysteroscopy. Also, no endocrine anomalies or autoimmune diseases were found, and both parents had normal karyotype. Sperm concentration was > 5 mill/ml. Only 6 women had 2 miscarriages (20%) and the remaining 24 women at least 3. They also had a PGS cycle with ≥ 60% of normal embryos.

Ages: 18 Years to 37 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bellver, MD, Principal Investigator — IVI Valencia
Locations (1):
- Ivi Valencia, Valencia, Valencia, Spain